CLINICAL TRIAL: NCT04012281
Title: International Post PCI FFR Registry for Prognostic Factors After Coronary Stenting
Brief Title: International Post PCI FFR Registry
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Tsuchiura Kyodo General Hospital (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other); Busan Veterans General Hospital (Unknown); Samsung Medical Center (Other); Sejong General Hospital (Other); Tokyo Medical University (Other); Gifu Heart Center (Other); Japanese Red Cross Kyoto Daini Hospital (Unknown); Inje University (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: 1906-152-1044
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Coronary Disease
Keywords: drug eluting stent; coronary atherosclerosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post PCI state: The study population of this study underwent percutaneous coronary intervention(PCI) with 2nd generation drug-eluting stent (DES) and measured fractional flow reserve after PCI
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — PCI was performed using 2nd generation DES

SUMMARY:
The prognostic factors after a percutaneous coronary intervention (PCI) have not been comprehensively investigated. The investigators sought to develop a risk model to predict future clinical events after PCI using contemporary coronary stents.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is a standard treatment strategy for coronary artery disease (CAD). With the presence of myocardial ischemia, PCI reduces the risks of death, myocardial infarction (MI) and revascularization compared to medical therapy. However, the risk of future clinical events still remain high and about 10% of patients experienced further cardiovascular events after PCI. There are several factors that are associated with these poor outcomes. Known patient-related risk factors are diabetes mellitus, chronic kidney disease, left ventricular dysfunction, previous MI and presentation with the acute coronary syndrome. Procedure-related factors, such as stent underexpension, malapposition, edge dissection, the number of the used stent and total stent length, are also related to poor prognosis after PCI. Recent studies reported that fractional flow reserve (FFR) after coronary stenting, or post PCI FFR, was associated with future clinical outcomes after PCI and low post PCI FFR value was associated with procedural factors. However, all of these risk factors were identified in individual studies there have been no studies that comprehensively evaluated these risk factors. Therefore, the investigators sought to investigate the risk predictors of future clinical events in patients after PCI and develop a risk model, incorporating clinical, angiographic, and physiologic factors, to predict the clinical events after PCI using contemporary coronary stents.

The study population of this study is from the International Post PCI FFR Registry, which included 4 different registries from Korea, China, and Japan. All patients in this registry are available with clinical, angiographic and physiologic data and used 2nd generation drug-eluting stent (DES) for PCI. The COE-PERSPECTIVE registry (NCT01873560) was designed to evaluate the clinical relevance of post PCI FFR from 9 hospitals in Korea and Japan and enrolled a total of 835 patients available post PCI FFR value after angiographically successful PCI between May 2013 and December 2016. The 3V-FFR-FRIENDS registry (NCT01621438) enrolled a total of 1,136 patients (3,298 vessels) who underwent 3-vessel FFR measurements from 12 centers in Korea, Japan, and China between November 2011 and March 2014. Among them, 266 patients with 337 vessels who measure post PCI FFR values were included in this international registry. The DKCRUSH VII registry (ChiCTR-PRCH-12001976) enrolled a total of 1,476 patients from 9 hospitals (5 hospitals in China, 2 hospitals in the United States, 1 hospital in Asia and 1 hospital in European country) between May 2012 and September 2013 to evaluate the prognostic value of post PCI FFR on patients' future outcome. For this international registry, 780 patients with 794 vessels from Nanjing First Hospital in China, who were available with whole clinical, angiographic and physiologic data, were included in this registry. Last, the Institutional registry of Tsuchiura Kyodo General Hospital, Ibaraki, Japan included 347 patients (357 vessels) who underwent PCI and final post-PCI FFR measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent PCI and post-PCI FFR measurements after angiographically successful stent implantation (residual stenosis < 20% by visual estimation)
* Patients who provided informed consent

Exclusion Criteria:

* Post-PCI TIMI flow of < 3
* Depressed left ventricular systolic function (ejection fraction < 30%)
* Culprit lesion for acute coronary syndrome
* Graft vessel
* Collateral feeder
* In-stent stenosis
* Primary myocardial or valvular heart disease
* Patients with life expectancy < 2 years.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as obstructive coronary artery disease and treated by 2nd generation DES and measured post PCI FFR after PCI.
Sampling Method: Non-Probability Sample
Enrollment: 2228 (Actual)
Dates: Start 2010-08-17 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Discrimination index of prediction model for target-vessel failure | 2 years after index procedure
  A risk model for target-vessel failure, incorporating clinical, angiographic, and additional physiologic predictors, will be developed using this cohort.
  Target vessel failure is a composite of cardiac death, clinically-driven target vessel-related myocardial infarction, and clinically-driven target vessel revascularization. The target vessel will be defined as the treated vessel with 2nd generation DES which was assessed by post stent fractional flow reserve.

SECONDARY OUTCOMES:
Independent predictors for target vessel failure | 2 years after index procedure
  Clinical, angiographic and physiologic covariables will be evaluated using machine learning for identifying the independent predictors (ex. random survival forest model).

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Director — Seoul National University Hospital; Joon Hyung Doh, MD, PhD, Principal Investigator — Inje University; Shao-Liang Chen, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University; Tsunekazu Kakuta, MD, PhD, Principal Investigator — Tsuchiura Kyodo General Hospital; Joo Myung Lee, MD, PhD, Principal Investigator — Samsung Medical Center

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Fearon WF, Nishi T, De Bruyne B, Boothroyd DB, Barbato E, Tonino P, Juni P, Pijls NHJ, Hlatky MA; FAME 2 Trial Investigators. Clinical Outcomes and Cost-Effectiveness of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention in Patients With Stable Coronary Artery Disease: Three-Year Follow-Up of the FAME 2 Trial (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation). Circulation. 2018 Jan 30;137(5):480-487. doi: 10.1161/CIRCULATIONAHA.117.031907. Epub 2017 Nov 2. PMID 29097450
- [Background] Hwang D, Lee JM, Lee HJ, Kim SH, Nam CW, Hahn JY, Shin ES, Matsuo A, Tanaka N, Matsuo H, Lee SY, Doh JH, Koo BK. Influence of target vessel on prognostic relevance of fractional flow reserve after coronary stenting. EuroIntervention. 2019 Aug 29;15(5):457-464. doi: 10.4244/EIJ-D-18-00913. PMID 30561367
- [Background] Li SJ, Ge Z, Kan J, Zhang JJ, Ye F, Kwan TW, Santoso T, Yang S, Sheiban I, Qian XS, Tian NL, Rab TS, Tao L, Chen SL. Cutoff Value and Long-Term Prediction of Clinical Events by FFR Measured Immediately After Implantation of a Drug-Eluting Stent in Patients With Coronary Artery Disease: 1- to 3-Year Results From the DKCRUSH VII Registry Study. JACC Cardiovasc Interv. 2017 May 22;10(10):986-995. doi: 10.1016/j.jcin.2017.02.012. Epub 2017 Apr 26. PMID 28456699
- [Background] Rimac G, Fearon WF, De Bruyne B, Ikeno F, Matsuo H, Piroth Z, Costerousse O, Bertrand OF. Clinical value of post-percutaneous coronary intervention fractional flow reserve value: A systematic review and meta-analysis. Am Heart J. 2017 Jan;183:1-9. doi: 10.1016/j.ahj.2016.10.005. Epub 2016 Oct 11. PMID 27979031
- [Background] van Zandvoort LJC, Masdjedi K, Witberg K, Ligthart J, Tovar Forero MN, Diletti R, Lemmert ME, Wilschut J, de Jaegere PPT, Boersma E, Zijlstra F, Van Mieghem NM, Daemen J. Explanation of Postprocedural Fractional Flow Reserve Below 0.85. Circ Cardiovasc Interv. 2019 Feb;12(2):e007030. doi: 10.1161/CIRCINTERVENTIONS.118.007030. PMID 30732469
- [Derived] Zhang J, Hwang D, Yang S, Kim CH, Lee JM, Nam CW, Shin ES, Doh JH, Hoshino M, Hamaya R, Kanaji Y, Murai T, Zhang JJ, Ye F, Li X, Ge Z, Chen SL, Kakuta T, Koo BK. Differential Prognostic Implications of Pre- and Post-Stent Fractional Flow Reserve in Patients Undergoing Percutaneous Coronary Intervention. Korean Circ J. 2022 Jan;52(1):47-59. doi: 10.4070/kcj.2021.0128. Epub 2021 Sep 24. PMID 34877828
- [Derived] Lee JM, Hwang D, Choi KH, Lee HJ, Song YB, Cho YK, Nam CW, Hahn JY, Shin ES, Doh JH, Hoshino M, Hamaya R, Kanaji Y, Murai T, Zhang JJ, Ye F, Li X, Ge Z, Chen SL, Kakuta T, Koo BK. Prognostic Impact of Residual Anatomic Disease Burden After Functionally Complete Revascularization. Circ Cardiovasc Interv. 2020 Sep;13(9):e009232. doi: 10.1161/CIRCINTERVENTIONS.120.009232. Epub 2020 Sep 8. PMID 32895005
- [Derived] Hwang D, Lee JM, Yang S, Chang M, Zhang J, Choi KH, Kim CH, Nam CW, Shin ES, Kwak JJ, Doh JH, Hoshino M, Hamaya R, Kanaji Y, Murai T, Zhang JJ, Ye F, Li X, Ge Z, Chen SL, Kakuta T, Koo BK. Role of Post-Stent Physiological Assessment in a Risk Prediction Model After Coronary Stent Implantation. JACC Cardiovasc Interv. 2020 Jul 27;13(14):1639-1650. doi: 10.1016/j.jcin.2020.04.041. PMID 32703590